CLINICAL TRIAL: NCT05693168
Title: Accuracy of Pulse Oximeter With Profound Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIBE01
Record Dates: First submitted 2022-12-27; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Comparison of ANNE Limb Sensor pulse oximetry measurements to blood gas analysis (Experimental)
  Interventions: Device: ANNE Limb Sensor

INTERVENTIONS:
Device: ANNE Limb Sensor — Pulse Oximeter

SUMMARY:
Clinical evaluation of the accuracy of SpO2 measurements with the ANNE Limb Sensor compared to blood gas analysis in healthy, adult subjects. Hypoxia is induced in patients to different and stable levels of SaO2 over the range of 70-100%.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, between the ages of 18 and 55 years.
* The subject is in good general health with no evidence of any medical problems
* The subject is fluent in both written and spoken English
* The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* Known history of heart disease, lung disease, kidney or liver disease
* Diagnosis of asthma, sleep apnea, or use of CPAP
* Subject has diabetes
* Subject has a clotting disorder
* The subject has a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation
* The subject has any other serious systemic illness
* Th subject is a current smoker
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators would interfere with the sensors working correctly
* The subject has a history of fainting or vasovagal response
* The subject has a history of sensitivity to local anesthesia
* The subject has a diagnosis of Raynaud's disease
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test)
* The subject is pregnant, lactating, or trying to get pregnant
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures
* The subject has any other condition, which in the opinion of the investigators would make them unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
ARMS of SpO2 Measurements with ANNE Limb compared to SaO2 | 1 hour
  Root mean square error between the function blood oxygen saturation (SpO2) provided by the device under test and the blood gas analysis of oxyhemoglobin saturation (SaO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Hypoxia Research Laboratory Department of Anesthesia and Perioperative Care University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No